CLINICAL TRIAL: NCT06603467
Title: Guided Versus Non-Guided Harvesting Technique of Soft Tissue Graft in Cairo Recession Type I Sites: a Randomized Clinical Trial
Brief Title: Guided Versus Non-Guided Harvesting Technique of Soft Tissue Graft in Cairo Recession Type I Sites
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, safinaz saleh mohamed saeed, lecturer in periodontology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #R-OMPDR-2-24-3097
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gingival Recessions
Keywords: gingival recessions
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): gingival recession will be covered with de-epithelialized free gingival graft harvested without guide
  Interventions: Procedure: non-guided de-epithelialized free gingival graft harvested
- group 2 (Active Comparator): gingival recession will be covered with de-epithelialized free gingival graft harvested with guide
  Interventions: Procedure: guided de-epithelialized free gingival graft harvested

INTERVENTIONS:
Procedure: non-guided de-epithelialized free gingival graft harvested — gingival recession will be covered with de-epithelialized free gingival graft harvested without guide
  Arms: group 1
Procedure: guided de-epithelialized free gingival graft harvested — gingival recession will be covered with de-epithelialized free gingival graft harvested with digital guide
  Arms: group 2

SUMMARY:
The goal of this clinical trial is to compare the healing pattern in the palate following harvesting of deepithelialized free gingival graft by two different harvesting techniques and to compare the recession coverage at the recipient sites.

. The main questions it aims to answer are:

• Does the harvesting technique will affect the healing pattern &the recipient site coverage in the treatment of gingival recession?

Participants will:

* Receive in the recession sites, in group 1 deepithelialized free gingival graft harvested without guide & group 2: will be covered with graft harvested with guide
* Visit the clinic twenty-four hours after surgery and weekly visits for 1 month, early wound healing at the sites of harvesting will be assessed
* The recession coverage will be assessed at 3& 6 months after surgery

DETAILED DESCRIPTION:
Background: Over the last few years, deepithelialized free gingival graft has become a gold standard treatment modality for increasing the width of keratinized gingiva, root coverage, alveolar ridge deficiencies management of peri-implant tissue abnormalities, and papillary loss. The procedure of harvesting the graft from the palate is often associated with the noteworthy challenge of procurement of the largest volume of tissue possible while minimizing associated trauma to anatomical structure, also special designs of the graft may be required. To meet these requirements and overcome the challenges, an innovative digitally designed guide for harvesting the graft is designed to allow ideally designed graft with minimal trauma to the tissue.

Aim: To compare the healing pattern in palate following harvesting of deepithelialized free gingival graft by two different harvesting techniques and to compare the recession coverage at the recipient sites.

Methodology: Twenty recession sites with RT1 Cairo classification will be recruited for this study. Sites were randomly divided into 2 treatment groups as follows: group 1 :10 sites will be covered with deepithelialized free gingival graft harvested without guide & group 2 :10 sites will be covered with CTG harvested with guide. Sites in both groups will be covered with laterally or coronally positioned flap. Twenty-four hours after surgery and weekly visits for 1 month, early wound healing at the sites of harvesting will be assessed using the Early Wound Healing Score (EHS) EHS. This score assessed clinical signs of re-epithelialization (CSR), clinical signs of hemostasis (CSH), and clinical signs of inflammation (CSI). Since complete wound epithelialization was the main outcome, the CSR score was weighted to be 60% of the total final score. Accordingly, a score of 0, 3, or 6 points was possible for the assessment of CSR, whereas scores of 0, 1, or 2 points were possible for CSH and CSI. Higher values indicated better healing. Accordingly, the score for ideal early wound healing was 10. Regarding soft tissue coverage, Gingival recession depth (GRD) & Gingival recession width (GRW) will be measured at baseline, 3 and 6 months after surgery. Also, each group will be subjected to intraoral scanning at baseline, 3 and 6 months after surgery to measure gingival thickness and level by superimposition of scanning files of different intervals to monitor the changes by software.

Statistical analysis will be done using IBM SPSS Statistics for Windows, version 23 (IBM Corp., Armonk, NY, USA). Intergroup analysis was done using Mann-Whitney test and intra-group analysis will be done using Kruskal-Wallis test for all the study parameters. Statistical significance will set at a p-value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Gingival recession sited classifies as Cairo type I
* must have a general health showing no contraindications for oral surgery,
* must be at least 20 years old.
* patients also had to have good oral hygiene before the treatment

Exclusion Criteria:

* signs or symptoms of bruxism or clenching i
* patients suffering from uncontrolled systemic conditions
* smoker
* pregnant or lactating

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Early Wound Healing Score (EHS) EHS | 6 month
  Early Wound Healing Score (EHS) EHS. This score assessed clinical signs of re-epithelialization (CSR), clinical signs of hemostasis (CSH), and clinical signs of inflammation (CSI). Since complete wound epithelialization was the main outcome, the CSR score was weighted to be 60% of the total final score. Accordingly, a score of 0, 3, or 6 points was possible for the assessment of CSR, whereas scores of 0, 1, or 2 points were possible for CSH and CSI. Higher values indicated better healing. Accordingly, the score for ideal early wound healing was 10

SECONDARY OUTCOMES:
Recession depth | 6 months
  Regarding soft tissue coverage, Gingival recession depth (GRD) from cementoenamel junction to Free gingival margin will be measured at baseline, 3 and 6 months after surgery.
gingival thickness | 6 months
  leach group will be subjected to intraoral scanning at baseline, 3 and 6 months after surgery to measure gingival thickness and level by superimposition of scanning files of different intervals to monitor the changes by software
recession width | 6 months
  measured at cementoenamel junction from mesial to distal line angel at baseline , 3 months & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: bassem nabil elfahl, lecturer in periodontology, Principal Investigator — Faculty of Dentistry, Tanta university
Locations (1):
- Faculty of Dentistry,Tanta university, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No